CLINICAL TRIAL: NCT01876758
Title: Cognitive Training for Memory Deficits Associated With Electroconvulsive Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #6599
Record Dates: First submitted 2013-06-03; First posted 2013-06-13 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Memory Deficits; Electroconvulsive Therapy
Keywords: ECT; Memory Training; Cognitive Remediation; Electroconvulsive Therapy; Treatment Resistant Depression; Depression; Geriatric Depression; Memory Loss; Cognitive Training
MeSH Terms: conditions — Memory Disorders; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Intervention: Memory Training (Experimental): Memory training before and after ECT
  Interventions: Behavioral: Cognitive Intervention: Memory Training
- Comparable general mental stimulation (Active Comparator): Puzzle games before and after ECT
  Interventions: Behavioral: Comparable general mental stimulation
- Treatment as Usual (No Intervention): No memory training or puzzle games, just the study evaluations

INTERVENTIONS:
Behavioral: Cognitive Intervention: Memory Training — Paper-and-pencil and computerized exercises pre- and post-ECT which may be helpful in recovering episodic memories and allow for the retention of learned strategies
  Arms: Cognitive Intervention: Memory Training
Behavioral: Comparable general mental stimulation — Active control will work on commercially available puzzle games at the same time prior and after ECT to determine if the developed memory training program is more effective than mere mental stimulation.
  Arms: Comparable general mental stimulation

SUMMARY:
Although electroconvulsive therapy (ECT) remains the most effective treatment for people with severe depression, patients may experience a significant degree of persistent and/or permanent memory problems following ECT. Many patients report the memory problems are the most disturbing and serious side effect of ECT, and that such effects impact their quality of life following treatment and their willingness to consent to further ECT needed to complete a treatment course or to maintain remission. New developments in the field of cognitive remediation have demonstrated the benefits of cognitive training to improve memory performance in various conditions, such as epilepsy. However, these strategies have never been applied to help patients regain memory after ECT. The investigators have designed and piloted a novel cognitive program specifically targeted to the cognitive effects of ECT, based upon a program tailored to people with seizure disorders, a group with memory problems very similar to people who undergo ECT. This Memory Training for ECT (Mem-ECT) is designed to help cognitive functions that may be compromised following ECT remain relatively preserved. In addition, the intervention attempts to help ECT patients quickly regain their general memory skills immediately following ECT. Recent results from our preliminary group of patients who underwent ECT and memory training at New York Presbyterian shows no overall decline in memory function following ECT. On the basis of these promising findings, the investigators propose a more rigorous and larger study to confirm whether this novel memory training program can help alleviate memory problems associated with ECT.

DETAILED DESCRIPTION:
The investigators propose to enroll 60 patients scheduled to undergo ECT over the course of 3 years. They will be randomly assigned to one of three research conditions (a) participants in Mem-ECT condition will receive memory training before and after their ECT course, (b) participants in the active control condition will work on commercially available puzzle games at the same times prior and after ECT to determine if the developed memory training program is more effective than mere mental stimulation, (c) participants in the "treatment as usual" will not work on the memory training or the puzzle games but just undergo the study evaluations. Participants will be evaluated a few days before ECT, within 2 weeks following ECT, and once again 2 months later. The evaluation will consist of interviews, mental skill testing, and measuring brain waves using an electroencephalograph (EEG) before ECT and 2 months after ECT (no EEG right after ECT). It is our hope that developing a safe and effective strategy to minimize the adverse memory side effects of ECT will make ECT a better and more easily tolerated treatment for patients with severe depression who need this therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder
* Inpatient at NYSPI or Presbyterian Hospital
* Scheduled to undergo right-unilateral electroconvulsive therapy in the next two weeks
* We do not require participants to be psychiatrically stable in terms of their symptoms. They only need to demonstrate capacity to consent and be willing to sit through 3 training sessions prior to ECT and 5 sessions post ECT

Exclusion Criteria:

* Significant auditory/visual impairment that would interfere with study procedures
* Lack of aptitude in English that may interfere with the administration of the tests
* Changes in the type of antidepressant during the course of ECT or 2 weeks post ECT
* Chart diagnosis of any other medical or neuropsychiatric illnesses known to impair brain function (e.g. mental retardation, traumatic brain injury, schizophrenia)
* History of ECT in past 2 months
* Mental status examination score below 40/57
* Current substance abuse (e.g. marijuana or crack), excluding nicotine and caffeine.
* Too agitated to sit through the required tests or training

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Columbia University Autobiographical Memory Interview-Short Form (AMI-SF) | 2 months after the last ECT session

SECONDARY OUTCOMES:
Goldberg Remote Memory Questionnaire | 2 months after the last ECT session
Hamilton Rating Scale for Depression-24 item | 2 months after the last ECT session

OTHER OUTCOMES:
Modified Mini-Mental State examination | 2 months after the last ECT session

CONTACTS AND LOCATIONS:
Overall Officials: Joan Prudic, MD, Principal Investigator — New York State Psychiatric Institute; Jimmy Choi, PsyD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Choi J, Lisanby SH, Medalia A, Prudic J. A conceptual introduction to cognitive remediation for memory deficits associated with right unilateral electroconvulsive therapy. J ECT. 2011 Dec;27(4):286-91. doi: 10.1097/YCT.0b013e31821d3ab3. PMID 22080239